CLINICAL TRIAL: NCT02587000
Title: Pilot Phase II, Randomized , and Control in Double Blind Placebo Effectiveness a 3 Months on Bleeding Fibroids Treatment With ULIPRISTAL ACETATE 10 mg/Day in Patients Suffering From Symptomatic Endometriosis
Brief Title: Adenomyosis and Ulipristal Acetate
Acronym: FRA-IIT-UPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P141201; 2014-004403-75 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-10-27 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2016-09

CONDITIONS: Adenomyosis
Keywords: adenomyosis; ulipristal acetate; sonography; Magnetic resonance imaging [MRI]; Pictorial Blood-loss Assessment Chart [PBAC]
MeSH Terms: conditions — Adenomyosis | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ulipristal acetate (Active Comparator): ESMYA® : 2 tablets of 5mg per day during 3 months, per os
  Interventions: Drug: Ulipristal acetate
- Placebo (Placebo Comparator): 2 tablets of 5mg per day during 3 months, per os
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulipristal acetate
  Other Names: ESMYA®
  Arms: Ulipristal acetate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Evaluation of efficiency of selective progesterone receptor modulators (SPRM) (Ulipristal acetate) on bleeding control and pain for patients with adenomyosis and wish to keep fertility.

DETAILED DESCRIPTION:
After inclusion according to criteria, 2 arms : placebo and Ulipristal acetate (UA) 10mg with randomisation, 1 patient with placebo for 3 patients with UA.

48 patients will be included in this trial. The end point will be the bleeding evaluated by Pictorial Blood-loss Assessment Chart (PBAC) score, the amenorrhea rate and the pain evaluated with visual analogic scale.

ELIGIBILITY:
Inclusion Criteria:

* Not postmenopausal women aged 30 to 50,
* Accepting to give consent informed in writing,
* Suffering from a symptomatic pelvic endometriosis (menorrhagia isolated or associated with pain)
* Diagnosis information, confirmed the adenomyosis (T2-weighted) MRI and/or transvaginal ultrasonography, in the 6 months preceding the inclusion-having a score of bleeding (PBAC) > 100 from J1 to J8 of the menstruation before the visit of inclusion,
* With an index of body mass (IMC) ≥18 and < 40,
* Using a reliable method of non-hormonal contraception (non-hormonal intrauterine device (IUDs), sexual abstinence, diaphragm, condoms or vasectomy by the partner, or having undergone a surgical sterilization),
* Willing and able to complete auto-questionnaires in french
* Had no difficulties to understand and communicate with the investigator and his representatives
* Affiliation to a social security or assign.

Exclusion Criteria:

* Patient with a hormonal oral contraceptive or with a hormonal intrauterine Device (IUD) contraceptive
* Patient with a history of surgery (other than a caesarean or a cervical conization) uterus, ablation endometrial or uterine artery embolization,
* With other than the endometriosis endometrial pathology,
* Suffering of myoma of type 0, 1, 2 or 3,
* Requiring a transfusion or having a ≤6g/dL hemoglobin
* Existence of systemic coagulation,
* History of thromboembolism
* Progestagen taking severe disorders in the month preceding the tour selection, and corticosteroids and aspirin in the previous week,
* Existence of Pathology renal, respiratory or cardiac severe or progressive,
* Having a disturbed liver function (defined by the aspartate aminotransferase (ASAT), Alanine Amino Transferase (ALAT), γGlutamylTranspeptidase, alkaline phosphatase or total bilirubin above 2 times the upper limit of normal),
* Existence or suspicion of malignancy,
* Considering pregnancy in the coming year,
* Pregnant patient or nursing
* Any clinical condition that the investigator considers incompatible with the conduct of the study in terms of acceptable security,
* Participation in courses at another clinical study
* Patient whose accession to the test procedures may be insufficient or for which a long term follow-up seems difficult to achieve
* Person under authorship or curators under safeguard of justice
* History of hypersensitivity to the ulipristal or any of the excipients of ESMYA ® 5 mg tablet.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a control uterine bleeding estimated by a score of Pictorial Blood-loss Assessment Chart (PABC) < 75 of 28 days to the discontinuation of the study (S13) | after 12 weeks of treatment

SECONDARY OUTCOMES:
Evolution of the PBAC score over 28 days compared to pre-treatment score (J1) | at week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment
Percentage of patients with uterine bleeding control estimated by a score of PBAC < 75 on 28 days | at week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evolution of the PBAC score calculated from the sum on the 28 days during the treatment period for the first day of control of uterine bleeding; | at Day 29
percentage of patients with amenorrhea estimated by a score of PBAC ≤2 on 28 days | to week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evolution of the PBAC score calculated from the sum on the 28 days during the treatment period for the first day of amenorrhea | for the first day of amenorrhea after the treatment
Evolution of pain through a Visual scale analogue between J1 and S5 (J29) S13 (J85) and M6 (S26 S28), | between day1 (before treatment) and week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evolution of analgesics using between each visit (number of days of treatment and the percentage of patients without analgesic over each period of 28 days of collection of the PBAC) and by bearing the information provided by the investigator | between day1 (before treatment) and week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evolution quality of life questionnaire with Uterine Fibroid Symptom and health related Quality of Life (UFS - QOL) questionnaire | between day1 (before treatment) and week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evolution of anemia by hemoglobin and ferritin concentration and coagulation by the CAW | between day1 (before treatment) and week5 (day29), week9 (day57), week13 (day85) and month6 (week26, week28) after starting of the treatment (Day1)
Evaluation of the adenomyosis by MRI or ultrasound transvaginal : existence/absence, focal length/diffuse, shallow/deep | Before the treatment and 6 months after beginning of the treatment
blood pressure and heart rate, respiratory rate | Before the treatment and up to 6 months after beginning of the treatment
Number of participants with adverse events and their grades as assessed by CTCAE v4.0 | Before the treatment and up to 6 months after beginning of the treatment
biological examinations: hemoglobin, ferritin, TCA. | Before the treatment and up to 6 months after beginning of the treatment
  Safety assessment
Frequency of flashes of heat, headache, thickening of the endometrium, uterine bleeding, ovarian cyst. | Before the treatment and up to 6 months after beginning of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hervé FERNANDEZ, MD, PhD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France